CLINICAL TRIAL: NCT04004598
Title: Golf Intervention for Veterans Exercise Study
Brief Title: Golf for Veterans Study
Acronym: GIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, George Salem, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS1500352
Record Dates: First submitted 2019-06-29; First posted 2019-07-02 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Exercise Training
Keywords: aging, exercise, golf, intervention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Phase I, Feasibility and Safety Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- golf training (Experimental): 12-week golf training program
  Interventions: Behavioral: golf training

INTERVENTIONS:
Behavioral: golf training — 12 weeks of training by Professional Golf Association professional

SUMMARY:
Aging is associated with physiological declines that could impair the ability to perform activities of daily living and thus impair the quality of life of older adults. Golf is an activity that challenges the balance, flexibility, and muscular systems of the golfer and could have important implications in addressing the physiological declines associated with aging. Golf also challenges the cognition of golfer and is typically performed in groups of 2-4 people; therefore, it could also have important implications for the cognitive and social health of older adults. This research will investigate the effects of an introductory, therapeutic golf program on the physiological, cognitive, and social well-being of older adults. Older adult military veterans (60-80 years) will participate in a 12-week introductory golf program specifically designed with older adults in mind. The intervention will be led by Professional Golf Association (PGA) professionals with experience in teaching older adults to golf. In order to assess the effectiveness of the intervention, the functional, physiological, and cognitive abilities of the participants will be evaluated as well as the overall well-being before and after the completion of the golf program. These adaptations will be evaluated through the use of biomechanical analysis, standardized older adult functional tests, validated surveys and questionnaires, and validated cognitive assessments.

DETAILED DESCRIPTION:
Implementing a 12-week introductory golf intervention designed for older military veterans will allow us to evaluate the usefulness of golf as a means to promote physical activity and well-being across the lifespan. Golf, while studied from a performance perspective, has not been studied as an intervention to promote physical activity and health in older adults. This study will contribute to our knowledge about the feasibility and effectiveness of golf as a means to promote wellness across the lifespan.

1.0 OBJECTIVES AND PURPOSE

OBJECTIVE 1: Quantify the changes in the functional, cognitive, and physiological abilities of older military veterans following a 12-week introductory golf intervention.

Hypothesis: Participants will demonstrate improved functional, cognitive and physiological abilities following the intervention.

OBJECTIVE 2: Quantify golf demands and performance including a biomechanical analysis of golf swings, putting and picking up a ball following a 12-week introductory golf intervention.

Hypothesis: The demands of the golf intervention will be similar to or greater than the demands during commonly utilized older adult balance and strengthening exercises.

OBJECTIVE 3: Evaluate the safety and feasibility of a 12-week introductory golf intervention.

Hypothesis 3A: Adverse events associated with the intervention will be minor and not more frequent than AE's associated with other activity programs in seniors.

Hypothesis 3B: Adherence to the program will greater than the adherence associated with other activity-intervention programs in seniors.

3.0 SELECTION AND WITHDRAWAL OF SUBJECTS

Participants will be recruited using physician referrals, flyers, and visits to community centers, military Veteran fitness/wellness classes, military Veteran organizations, and military Veteran housing facilities in the Greater Los Angeles area. Once identified, the participants will go through a two-part screening process that includes a phone interview and clearance from their primary care physician. The phone screen includes the Telephone Memory Impairment Screen and a series of questions pertaining to the inclusion and exclusion criteria. Participants that pass the phone screen will be then required to receive clearance from their primary care physician prior to enrollment in the study. At the baseline testing session, additional details of the study will be explained to the participants, and consent obtained by an experienced researcher.

4.0 RISK ANALYSIS The functional assessments include activities that are regularly conducted throughout the day and have been utilized regularly as part of common clinical practice for assessing functional abilities. In more challenging activities, the participants will be appropriately spotted to ensure safety during the test.

The potential risks are as follows:

Functional Assessment: Fatigue (very minimal risk) - Rest will be provided as needed for the participants.

Muscle soreness (minimal risk) - This is no greater than performing normal activities of daily living.

Joint or muscle injury (minimal risk) - This is no greater than performing normal activities of daily living.

Risk of falling (minimal risk) - On the more challenging tasks, participants will be spotted.

Cognitive Assessment: Questionnaires (minimal risk) - Participants will be given the option to skip or stop answering any questions that make them uncomfortable.

Golf Intervention: Joint or muscle injury (minimal risk) - The participants will be gradually introduced to the activities associated with the sport of golf. Each golf session will include a sport specific warm-up and exercises that prepare the participants for the daily activities. Additionally, the golfers will be supervised by a PGA Professional who specializes in instructing older adults.

Fatigue (very minimal risk) - Participants will also be allowed rest as needed.

Adverse Events: Any unanticipated problem will be recorded via an incident report. Protocols for the USC MBRL have been developed. Any serious adverse event will be reported to the Institutional Review Board at the USC Health Science Campus using the flow chart below.

Continual Safety Monitoring: Researchers will have weekly meetings with the PGA instructors to keep informed about the intervention and participant safety. Additionally, each week, research associates will check in with participants according to the Problem Reports and Tracking Problems Protocol.

5.0 CLINICAL/LABORATORY EVALUATIONS AND STUDY CALENDAR

Duration and Locations: The study from consent enrollment to final data collection will occur over a 16-week period. The study consists of two data collection visits to the Jacquelin Perry Musculoskeletal Biomechanics Research Laboratory (MBRL) in the Division of Biokinesiology and Physical Therapy located on the University of Southern California Health Science Campus and two data collection visits to a private room located at the West Los Angeles Veterans Administration Hospital (WLAVA). Day 1 (USC) and Day 2 (WLAVA) will occur following the consent enrollment (before training) and Day 3 (USC) and Day 4 (WLAVA) will occur following the completion of the training program.

Biomechanical Analysis at USC (minimal risk): Laboratory kinematics and kinetics will be collecting using an 11-camera digital motion capture system (Qualysis, AB, Gothenberg, Sweden). 14 mm reflective markers will be used to define body segments and track motion during the trials. The trunk will be modeled as 2 rigid segments: pelvic and spine segments. The lower extremity will be modeled as 3 rigid segments: thigh, shank and foot.

Day 1 Tasks (minimal risk): Data collection will last approximately 2 hours and will include previously validated functional assessments.

Height, mass, resting heart rate, resting blood pressure and body fat percentage via Bioelectrical Impedance Analysis 6 minute walk test Hip muscle performance Gait analysis Modified Tandem Quiet Standing Balance confidence: Activities Specific Balance Confidence (ABC) Scale Participants will be given a Golf History Form to complete at home and return on Day 2

Day 2 Tasks (minimal risk): Data collection will last approximately 1.5 hours and will include previously validated cognitive and self-efficacy assessments as well functional measures.

Participants will turn in their Golf History Form Self-reported health-related quality of life as assessed by the RAND 12-item Health Survey Surveys from the Midlife in the United States Survey (MIDUS) study assessing Positive and Negative affect, Social Well-Being, and Sense of Control Cognition as assessed by the NIH Toolbox for cognition Physical activity habits will be assessed via a questionnaire developed by the Postmenopausal Estrogen/Progestins Intervention (PEPI) Study and a physical activity free recall Episodic verbal learning and memory as assessed by the California Verbal Learning Test Senior Fitness Test: 30-second chair stand and 8-foot-up-and-go test

Day 3 Tasks (minimal risk): Data collection will last approximately 3 hours and will include all tasks performed on Day 1 plus a biomechanical analysis of golf-related demands (see below).

Golf swings, chips and putts that are common to recreational golf players. Participants will perform up to 5-10 trials of each swing type.

Picking up and setting down a golf ball. Subjects will perform up to 5-10 trials of each strategy.

Exit questionnaire about golf training program

Day 4 Tasks (minimal risk): Data collection will last approximately 2 hours and will include all tasks performed on Day 2.

Six months after the completion of the study, participants will receive a telephone call to follow-up on their current golf playing habits following the 12-week program.

Golf Training Visits: Participants will participate in golf training programs at the Heroes Golf Course on the WLAVA campus. Participants will be divided into groups of 2-4 golfers and will meet with a PGA Professional two times per week for 12 weeks. Training sessions will last 1-2 hours. The program is specifically designed for older adults not currently playing golf. The first set of sessions will include introduction to the different forms of the golf swing beginning with partial swings and then gradually progressing to a full swing. Swing modifications will be provided on an individual basis to address needs of the participant. Golf play will begin on holes that are flatter and close to the clubhouse and will begin by only playing 1-2 holes. The golfers will then be appropriately progressed to longer golf play as the PGA Professional feels it is appropriate. All equipment and fees will be included and there will be no cost to the participants.

Tasks (minimal risk):

Warm-up: Each training session will begin with a sport specific warm-up that prepares the participants for the activities of the day.

Supplementary Exercises: Additional strengthening and flexibility exercises will be included in training sessions to prepare the participants for golf-related activities.

Golf swings and putting: These movements will be introduced in a progressive nature beginning with partial swings of the least forceful swing type and eventually progressing to the more forceful swings (drives). Swings with the following equipment will be included: putters, pitching or sand wedges, irons, and woods.

Picking up a ball: The participants will be introduced to techniques to picking up a golf ball which will be individualized to the needs of the participants based off current research in the MBRL (HS-15-00038).

Walking: Participants will gradually increase walking distance. Practice will begin on flat holes and will progress to holes with more challenging terrain.

Golf play: Participants will be gradually introduced to regular golf play beginning with play on a single, low difficulty hole and progressing to multiple holes. Skill difficulty will also be gradually increased.

During the intervention, walking distance will be tracked via fitness trackers. Golf performance will be tracked as well.

6.0 DATA COLLECTION AND MONITORING

Data will be stored securely in the MBRL, CHP, room G9. Electronic data will be stored on a password protected computer. Hard copies of data will be stored in a locking file cabinet. No subject identifiers will be collected.

7.0 STATISTICAL ANALYSIS 7.1 PRIMARY DEPENDENT VARIABLES

7.1.1 Segment/joint angular positions, velocities, and accelerations 7.1.2 Joint torques 7.1.3 COP dynamics 7.1.4 Static and dynamic balance 7.1.5 Hip Muscle Performance 7.1.6 Gait speed 7.1.7 Gait spatiotemporal characteristics 7.1.8 Cognitive-Motor Dual Task Performance 7.1.9 Activities Specific Balance Confidence 7.1.10 Senior Fitness Test 7.1.11 Self-Rated Health 7.1.12 Verbal memory recall 7.1.13 Positive and Negative affect 7.1.14 Personal Mastery 7.1.15 Perceived Constraints 7.1.16 Social Contribution 7.1.17 Cognition Fluid Composition Score

7.2 POWER ANALYSIS

To date, this study has not been conducted and thus no preliminary data was available for a power analysis. 12 subjects are requested to ensure for adequate sample size and account for study attrition, based on other exercise intervention studies in older adults.

7.3 STATISTICAL ANALYSIS Pre-Post comparisons will be made.

8.0 REGISTRATION GUIDELINE

Following confirmation of the inclusion and exclusion criteria, all potential participants will be consented before enrollment in the study. Study research associates have undergone CITI Training for human subjects' research. In order to participate in the study, participants must be English speaking and have the ability to follow instructions (as assessed by the Telephone Memory Impairment Screen); therefore, there is no need of a legally authorized representative during the consent process. Participants will be consented using a USC Informed Consent form after being explained the details of the study and allowing for adequate time to ask questions and make a decision.

ELIGIBILITY:
INCLUSION CRITERIA

* Older Military Veterans: 60-80 years old
* The ability to stand independently without external support
* No previous golf experience
* Played ≤1 time in the last month
* Played ≤3 times in the last 6 months
* English Speaking

EXCLUSION CRITERIA

* Dementia and Alzheimers Disease assessed via the Telephone Memory Impairment Screen
* Symptomatic cardiovascular disease, active angina, uncontrolled hypertension (SBP>160 or DBP>90, high resting pulse HR>90), symptomatic orthostatic hypotension
* Unstable asthma, exacerbated COPD
* Rheumatoid arthritis, unstable ankle, knee, hip, shoulder or wrist joints
* History of injury or orthopedic operation within the last 6 months
* Movement disorders (Parkinson's disease or other neurological disorders), stroke, hemiparesis or paraparesis
* Peripheral neuropathies, severe vision or hearing problems, or metastatic cancer
* Individuals with vestibular, visual, musculosketelal, orthopedic and/or neurological disorders known to impair balance

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Change in Gait speed | baseline and after 12 weeks
  change in walking speed

SECONDARY OUTCOMES:
Change in Strength | baseline and after 12 weeks
  change in dynamic and static strength

OTHER OUTCOMES:
Change in cognition | baseline and after 12 weeks
  Change in National Institute of Health Toolbox Fluid Cognition Composite Score Fully-corrected T Score metric normative mean of 50 and an SD of 10. Range is 0-100. Higher scores reflect better outcomes.
  The Fluid Cognition Composite Score is comprised of 5 subscales Dimensional Change Card Sort Test (measures executive function) Flanker Inhibitory Control and Attention Test measures attention and executive function Picture Sequence Memory Test (measures episodic memory) List Sorting Working Memory Test (measures working memory) Pattern Comparison Test (measures processing speed) Composite score is derived by averaging the standard scores of each of the five subscales. All subscales scores the same T-score metric
Change in balance | baseline and after 12 weeks
  change in dynamic and static balance

CONTACTS AND LOCATIONS:
Overall Officials: George J Salem, PhD, Principal Investigator — University of Southern California; Steve Castle, MD, Study Director — West Los Angeles Veterans Administration
Locations (2):
- United States (2):
  - University Southern California, Los Angeles, California
  - West Los Angeles Veterans Administration, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao KL, Hui-Chan CW, Tsang WW. Golfers have better balance control and confidence than healthy controls. Eur J Appl Physiol. 2011 Nov;111(11):2805-12. doi: 10.1007/s00421-011-1910-7. Epub 2011 Mar 17. PMID 21416145
- [Background] Tsang WW, Hui-Chan CW. Effects of exercise on joint sense and balance in elderly men: Tai Chi versus golf. Med Sci Sports Exerc. 2004 Apr;36(4):658-67. doi: 10.1249/01.mss.0000122077.87090.2e. PMID 15064594
- [Background] Tsang WW, Hui-Chan CW. Static and dynamic balance control in older golfers. J Aging Phys Act. 2010 Jan;18(1):1-13. doi: 10.1123/japa.18.1.1. PMID 20181990
- [Background] Hoerster KD, Lehavot K, Simpson T, McFall M, Reiber G, Nelson KM. Health and health behavior differences: U.S. Military, veteran, and civilian men. Am J Prev Med. 2012 Nov;43(5):483-9. doi: 10.1016/j.amepre.2012.07.029. PMID 23079170
- [Background] Littman AJ, Forsberg CW, Koepsell TD. Physical activity in a national sample of veterans. Med Sci Sports Exerc. 2009 May;41(5):1006-13. doi: 10.1249/MSS.0b013e3181943826. PMID 19346987
- [Background] Bouaziz W, Lang PO, Schmitt E, Kaltenbach G, Geny B, Vogel T. Health benefits of multicomponent training programmes in seniors: a systematic review. Int J Clin Pract. 2016 Jul;70(7):520-36. doi: 10.1111/ijcp.12822. Epub 2016 Jun 13. PMID 27291143
- [Background] Broman G, Johnsson L, Kaijser L. Golf: a high intensity interval activity for elderly men. Aging Clin Exp Res. 2004 Oct;16(5):375-81. doi: 10.1007/BF03324567. PMID 15636463
- [Background] Parkkari J, Natri A, Kannus P, Manttari A, Laukkanen R, Haapasalo H, Nenonen A, Pasanen M, Oja P, Vuori I. A controlled trial of the health benefits of regular walking on a golf course. Am J Med. 2000 Aug 1;109(2):102-8. doi: 10.1016/s0002-9343(00)00455-1. PMID 10967150
- [Background] Foxworth JL, Millar AL, Long BL, Way M, Vellucci MW, Vogler JD. Hip joint torques during the golf swing of young and senior healthy males. J Orthop Sports Phys Ther. 2013 Sep;43(9):660-5. doi: 10.2519/jospt.2013.4417. PMID 23886577
- [Background] Ball KA, Best RJ. Different centre of pressure patterns within the golf stroke I: Cluster analysis. J Sports Sci. 2007 May;25(7):757-70. doi: 10.1080/02640410600874971. PMID 17454544
- [Background] Bezzola L, Merillat S, Jancke L. The effect of leisure activity golf practice on motor imagery: an fMRI study in middle adulthood. Front Hum Neurosci. 2012 Mar 29;6:67. doi: 10.3389/fnhum.2012.00067. eCollection 2012. PMID 22479243
- [Background] Bezzola L, Merillat S, Gaser C, Jancke L. Training-induced neural plasticity in golf novices. J Neurosci. 2011 Aug 31;31(35):12444-8. doi: 10.1523/JNEUROSCI.1996-11.2011. PMID 21880905
- [Background] Murray AD, Daines L, Archibald D, Hawkes RA, Schiphorst C, Kelly P, Grant L, Mutrie N. The relationships between golf and health: a scoping review. Br J Sports Med. 2017 Jan;51(1):12-19. doi: 10.1136/bjsports-2016-096625. Epub 2016 Oct 3. PMID 27697939